CLINICAL TRIAL: NCT03385174
Title: Carbon Monoxide Headache Triggering Properties as Well as Effects on the Brain's Vessels and Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Hashmat Ghanizada, Principal investigator, Danish Headache Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-17016387
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Headache Disorders
MeSH Terms: conditions — Headache Disorders | interventions — Carbon Monoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carbon monoxide (Other): Each participant receives CO inhalation
  Interventions: Other: Carbon monoxide

INTERVENTIONS:
Other: Carbon monoxide — Carbon monoxide inhalation

SUMMARY:
Studying Carbon monoxide effects on brain vessels in healthy volunteers with magnetic resonance imaging.

DETAILED DESCRIPTION:
In this study we will systematically investigate the headache-releasing properties of carbon monoxide as well as measure the effect of carbon monoxide on mean blood flow rate in the brain's large vessel with magnetic resonance imaging. These studies are important for understanding and further investigating the carbon monoxide's headache-releasing effect in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18-50
* 50-100 kg

Exclusion Criteria:

* Tension type headache more than 5 dage /month
* Other primary headaches
* Daily medication except contraceptives
* Drug taken within 4 times the halflife for the specific drug except contraceptives
* Pregnant or lactating women
* Exposure to radiation within the last year
* Headache within the last 24 hours before start of trial
* Hypertension
* Hypotension
* Respiratory or cardiac disease
* Smoking
* Primary relatives with current or previous migraine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Changes in brain blood vessels diameters after a short CO inhalation | 30 minutes
  To investigate changes in the circumference of intra- and extracerebral blood vessels after inhalation of carbon monoxide using magnetic resonance angiography (MRA).

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark